CLINICAL TRIAL: NCT05102422
Title: Quantitative Electroencephalogram and Bispectral Index Brain Mapping During Propofol vs Sevoflurane General Anesthesia A Randomized Comparative Trial
Brief Title: Quantitative Electroencephalogram and Bispectral Index Brain Mapping During Propofol vs Sevoflurane General Anesthesia
Status: Completed | Type: Observational
Sponsor: Pierre Pandin (Other)
Responsible Party: Sponsor-Investigator, Pierre Pandin, MD, Erasme University Hospital
Organization: Erasme University Hospital (Other)
Other Study IDs: brainmap
Record Dates: First submitted 2021-10-04; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Neurophysiology
Keywords: General anesthetics; Bispectral index; Quantitative electroencephalography; Monitoring
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1-Propofol: Induction and maintenance of general anesthesia using the intravenous anesthetic.
  Every patient received an intravenous bolus of 0,2 μg.kg-1 sufentanil, and the propofol (P) infusion was started using target-controlled infusion (TCI - Schnider's pharmacokinetic/pharmacodynamic data set); targeting the effect-concentration of 3 µg.ml-1. The effect concentration was gradually increased by 1µg.ml-1 every 2 to 3 minutes until loss of consciousness occurred. 0.1 mg.kg-1 of iv cisatracurium was given to prepare definitive intubation. The P effect-concentration were increased of 1 µg.ml-1 until test laryngoscope was successful and oro-tracheal intubation was performed.
  The effect concentration of propofol is reduced to 3 to 4 µg.ml-1 while awaiting the surgical incision. It is then left to the discretion of the anesthetist to add either an iv bolus of sufentanil (0.1 μg.kg-1) and/or an iv bolus of cisatracurium (0.1 mg.kg-1) only if necessary, in the clinical judgment of the practitioner.
  Interventions: Drug: Propofol 1 % Injectable Suspension
- 2-Sevoflurane: Induction and maintenance of general anesthesia using the inhaled anesthetic sevoflurane.
  Every patient received an intravenous (iv) bolus of 0,2 μg.kg-1 sufentanil, then sevoflurane (S) is started at one minimal alveolar concentration (2% in 50% oxygen) during mask assisted ventilation. The S concentration is gradually incremented by 2% until the LOC when the mask ventilation became fully assisted. 0.1 mg.kg-1 of iv cisatracurium was given to prepare definitive intubation. The S end-tidal concentration were increased of 1% until the test laryngoscope was successful and oro-tracheal intubation was performed. The end-tidal concentration of sevoflurane is reduced to one MAC while awaiting the surgical incision.
  After surgical incision, it is left to the discretion of the anesthetist to add either an iv bolus of sufentanil (0.1 μg.kg-1) and/or an iv bolus of cisatracurium (0.1 mg.kg-1) only if necessary, in the clinical judgment of the practitioner.
  Interventions: Drug: Sevoflurane inhalant product

INTERVENTIONS:
Drug: Propofol 1 % Injectable Suspension — Induction and maintenance of general anesthesia using the intravenous anesthetic
  Other Names: Diprivan
  Groups: 1-Propofol
Drug: Sevoflurane inhalant product — Induction and maintenance of general anesthesia using the inhaled anesthetic sevoflurane
  Other Names: Sevorane
  Groups: 2-Sevoflurane

SUMMARY:
General anesthesia interferes with the whole cerebral cortex at different levels. The goal was to investigate the impact of general anesthesia on different regions of the cerebral cortex by recording the brain's electrophysiological activity using QEEG and BIS during general anesthesia for 40 patients undergoing orthopedic surgeries under general anesthesia to see whether our hypothesis, that there is a topographically-dependent impact of general anesthesia on different regions of the cerebral cortex, is valid or not. The patients were randomly divided into 2 groups of 20 patients to compare the effect on the brain function monitoring (QEEG vs BIS) of the intravenous anesthesia (propofol) with the halogenated anesthesia (sevoflurane). And finally, we compared the two brain function monitoring techniques, BIS and QEEG.

DETAILED DESCRIPTION:
After approval by the ethics committee, every patient signed a consent form to participate in this observational prospective open-label randomized study. We identified potential participants in the anesthesia pre-admission unit who presented to be seen by an anesthesiologist before their intervention. Details of eligibility criteria described later.

According to the international 10-20 reference system, 4 silver cup electrodes were placed on the left prefrontal (Fp1), parietal (P7), temporal (T7), and occipital (O1) points with the vertex (Cz) as a common reference after an adequate preparation of each scalp skin location using a micro-abrasive paste and degreasing using ethyl ether. The cup electrodes were placed and fixed on the skin with adhesive paste . After a similar skin preparation, an adult adhesive EKG surface electrode was secured to the patient's forehead as a cephalic ground electrode. Thus, by using 6 electrodes, we obtain a 4 channels set-up (prefrontal Fp1-CZ, parietal P7-Cz, temporal T7-Cz, and occipital O1-Cz) with a common vertex reference.

Each of the six electrodes of the montage are respectively connected to one special Y adapter including a double connection to be attached at the same time to the EEG amplifier, for the QEEG recording, and to the A1000™ Aspect Medical System™ amplifier, for the BIS recording. After the initial test of the electrode impedance (<5000 Ω), this last one was automatically checked all along the investigation to maintain the electrodes impedance below the same threshold. Regarding the QEEG, the low- and the high-frequency filters were set at 0.5 and 30 Hertz (Hz), respectively. EEG five seconds long epochs were sampled every 30 seconds for further analysis in the three respective domains (frequency, time, and power) in each EEG channel. Concerning the BIS monitoring, the EEG low- and high-frequency filters were set similarly to the QEEG whereas EEG sampling corresponds to 5-second segments of traces without smoothing, every 30 seconds. Finally, the BIS and its ancillary parameters simultaneously calculated in each channel, were extracted every 30 seconds. The selection of parameters for the QEEG analysis included Spectral Edge Frequency (SEF), Median EEG Frequency (MEF), Burst Suppression Ratio (BSR) and Total Spectral Power (TSP). Regarding the bispectral EEG analysis, the only parameter was the BIS itself. Thus, each parameter value is obtained for each channel during EEG and BIS sampling. Finally, for clinical monitoring, heart rate (HR), mean arterial pressure (MAP) and pulse oximetry (Sa02) were considered.

After the standard clinical monitoring placement (ECG, non-invasive arterial pressure cuff and ear/finger pulse oximetry device) and a peripheral venous catheter insertion connected to an infusion line, the non-premedicated patients were preoxygenated with a facial mask with 100% oxygen. Capnography via nasal cannula were initially applied and monitored prior to the anesthetic induction and replaced by the manual ventilation system when needed during the general anesthesia (GA) effect occurrence. First, every patient received an intravenous (iv) bolus of 0,2 μg.kg-1 sufentanil. After that, in the group 1 the propofol (P) infusion was started using target-controlled infusion (TCI) with a Total IntraVenous Anesthesia (TIVA) pump (Schnider's pharmacokinetic/pharmacodynamic data set); targeting the effect-concentration of 3µg.ml-1. From then on, the effect concentration was gradually increased by 1µg.ml-1 every two to three minutes until loss of consciousness (LOC as loss of verbal contact, spontaneous ventilation, corneal reflex, and ciliary reflex) occurred. At this point the effect concentration level of propofol upon loss of consciousness (PROPLOC) is recorded. At the same time, in group 2, sevoflurane (S) is started at one minimal alveolar concentration (2% in 50% oxygen) during mask assisted ventilation. Then, in a similar manner to group 1, the S concentration is gradually incremented by 2% until the LOC when the mask ventilation became fully assisted. The corresponding S effect-concentration (SEVOLOC) was also noted. Subsequently, the LOC confirmed, after an interval of 1 to 2 minutes, a first laryngoscopy was performed to test the possibility of intubation of the patients. In case of adequate intubation conditions (no physical or hemodynamical reaction to laryngoscopy and/or normal airway compliance), 0.1 mg.kg-1 of iv cisatracurium was given to prepare definitive intubation. When the patients did not encounter correct intubation conditions (first laryngoscopy failure), the P effect-concentration and the S end-tidal concentration were respectively increased of 1µg.ml-1 and 1% until the test laryngoscope was successful. After intravenous cisatracurium administration, manually assisted ventilation was conducted for 3 minutes in a way to have the partial pressure of end-tidal carbon dioxide (etCO2) between 32-35 mmHg. Intubation followed and intermittent positive pressure ventilation was used maintaining the same values of etCO2. The corresponding drug concentrations of propofol at intubation (PROPIntub) and sevoflurane at intubation (SEVOIntub) were recorded. From the moment the patient is mechanically ventilated, the effect concentration of propofol and the end-tidal concentration of sevoflurane are reduced to 3 to 4 µg.ml-1 and one minimal alveolar concentration (MAC) respectively while awaiting the surgical incision. Then, during the following 15-minute period of data collection no external stimuli were permitted on or around the patient. This pharmacological steady-state period was considered for the comparative topographic analysis between the different electrode categories regarding the general anesthesia effect on the brain. Therefore, the intraoperative period extends from the surgical incision to the end of the surgery. During this period, it is left to the discretion of the anesthetist to add either an iv bolus of sufentanil (0.1 μg.kg-1) and/or an iv bolus of cisatracurium (0.1 mg.kg-1) only if necessary, in the clinical judgment of the practitioner. To note, the parametric values of the QEEG and BIS were not considered to guide the anesthesia throughout the investigation. The postoperative period begins after the end of surgery when the anesthesia is stopped and lasts until the patient is awake and calm, ready to leave the operating room after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (BMI<27)
* American Society of Anesthesiologists (ASA) I and II (classification of the American Society of Anesthesiologists) adult patients
* Undergoing an orthopedic surgery
* Under general anesthesia
* Supine position

Exclusion Criteria:

* History of allergy, intolerance, or reaction to propofol or to sufentanil or hypersensitivity to either drug
* History of allergy, intolerance or reaction to sevoflurane or hypersensitivity to this drug
* History of malignant hyperthermia to sevoflurane or other halogenated gaz
* History of allergy, intolerance, or reaction to cisatracurium or hypersensitivity to this drug
* Any history of neurologic, neurovascular, neurosurgical, or psychiatric active pathology within past 6 months
* History of allergy to egg, soy, or lecithin
* Uncontrolled arterial hypertension
* Unstable cardiac status (life-threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction)
* Concomitant use of opioids, b-receptor antagonist, a2-receptor agonist or calcium channel blocker
* Currently receiving pharmacological agents for hypertension or cardiac disease
* Currently receiving or has received digoxin within the past 3 months BMI >28 kg m²
* Active, uncontrolled gastro-oesophageal reflux - an aspiration risk
* Current (or within past 3 months) history of apnea requiring an apnea monitor
* Craniofacial anomaly, which could make it difficult to effectively establish a mask airway for positive pressure ventilation if needed
* Active, current respiratory issues different from the baseline status (pneumonia, exacerbation of asthma, bronchiolitis, respiratory syncytial virus)
* Refusal of insertion of intravenous catheter while awake
* Patient refusal to participate in the study
* Cerebro-motor retardation / Mental disability / Psychological dependence / Legal guardianship

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an orthopedic surgery to be operated in Erasme hospital, Belgium
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-08-21 (Actual); Primary Completion 2009-12-15 (Actual); Study Completion 2009-12-15 (Actual)

PRIMARY OUTCOMES:
Frequency domain analysis QEEG | intraoperatively
  Spectral Edge Frequency (Hz) and Median EEG Frequency (Hz) in the four cerebral cortical territories considered (PreFrontal Fp1; Temporal T7; Parietal and Occipital)
Time domain analysis QEEG | intraoperatively
  BSR (Burst Suppression Ratio) in % in the four cerebral cortical territories considered
Power domain analysis QEEG | intraoperatively
  Total Spectral Power (TSP) in the four cerebral cortical territories considered
BIS | intraoperatively
  BIS recordings in the four cerebral cortical territories studied

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Pandin, MD, Study Director — Erasme University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] John ER, Prichep LS, Kox W, Valdes-Sosa P, Bosch-Bayard J, Aubert E, Tom M, di Michele F, Gugino LD. Invariant reversible QEEG effects of anesthetics. Conscious Cogn. 2001 Jun;10(2):165-83. doi: 10.1006/ccog.2001.0507. PMID 11414713
- [Background] John ER, Prichep LS. The anesthetic cascade: a theory of how anesthesia suppresses consciousness. Anesthesiology. 2005 Feb;102(2):447-71. doi: 10.1097/00000542-200502000-00030. No abstract available. PMID 15681963
- [Background] Cimenser A, Purdon PL, Pierce ET, Walsh JL, Salazar-Gomez AF, Harrell PG, Tavares-Stoeckel C, Habeeb K, Brown EN. Tracking brain states under general anesthesia by using global coherence analysis. Proc Natl Acad Sci U S A. 2011 May 24;108(21):8832-7. doi: 10.1073/pnas.1017041108. Epub 2011 May 9. PMID 21555565
- [Background] Hudetz AG. General anesthesia and human brain connectivity. Brain Connect. 2012;2(6):291-302. doi: 10.1089/brain.2012.0107. PMID 23153273
- [Background] Pandin P, Van Cutsem N, Tuna T, D'hollander A. Bispectral index is a topographically dependent variable in patients receiving propofol anaesthesia. Br J Anaesth. 2006 Nov;97(5):676-80. doi: 10.1093/bja/ael235. Epub 2006 Aug 23. PMID 16928697